CLINICAL TRIAL: NCT00235469
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Assess the Efficacy and Safety OF 200, 400, AND 600 mg/Day SPM 927 in Subjects With Painful Distal Diabetic Neuropathy
Brief Title: A Trial to Assess the Efficacy and Safety of SPM 927 in Subjects With Painful Distal Diabetic Neuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP0742
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2010-02

CONDITIONS: Diabetic Neuropathy
Keywords: PAINFUL DISTAL DIABETIC NEUROPATHY
MeSH Terms: conditions — Diabetic Neuropathies | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

INTERVENTIONS:
Drug: SPM 927

SUMMARY:
This phase 2b trial is being conducted at approximately 60 sites in the US to investigate whether lacosamide (SPM 927) at different doses reduces pain in subjects with diabetic neuropathy. Approximately 360 subjects will be randomized to placebo or one of three doses of lacosamide. To qualify for this trial, subjects with symptoms of painful distal diabetic neuropathy ranging in duration from 6 months to 5 years must have an average pain intensity of ≥4 on an 11-point Likert scale (0-10 scale) during the 7 day period prior to start of treatment.

To determine what effect lacosamide has on diabetic neuropathic pain, subjects will use a diary to record their daily pain intensity (morning and evening), pain interference with sleep (morning) and activity (evening). Use of rescue medication (acetaminophen) and subjects' quality of life will be investigated. In addition, safety and tolerability of the different doses of lacosamide will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Painful distal diabetic neuropathy

Exclusion Criteria:

* Must have an average pain intensity of ≥ 4 on an 11-point Likert scale

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2004-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To investigate the efficacy of 200, 400, and 600 mg/day of lacosamide compared with placebo in reducing pain in subjects with painful distal diabetic neuropathy.

SECONDARY OUTCOMES:
To investigate the effect of lacosamide on subjects' perception of pain, sleep, activity, quality of life, as well as to investigate the pharmacokinetics and safety of lacosamide.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, RTP, North Carolina, United States

REFERENCES:
- [Result] Wymer JP, Simpson J, Sen D, Bongardt S; Lacosamide SP742 Study Group. Efficacy and safety of lacosamide in diabetic neuropathic pain: an 18-week double-blind placebo-controlled trial of fixed-dose regimens. Clin J Pain. 2009 Jun;25(5):376-85. doi: 10.1097/AJP.0b013e318196d2b6. PMID 19454870